CLINICAL TRIAL: NCT03590743
Title: A Phase IV, Randomized, Double Blind Study Evaluating the Safety and Efficacy of Apixaban in Subjects With Calf Vein Thrombosis
Brief Title: Calf Deep Vein Thrombosis Treatment Trial
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of participant enrollment
Sponsor: Mayo Clinic (Other)
Collaborators: Bristol-Myers Squibb (Industry); Pfizer (Industry)
Responsible Party: Principal Investigator, Robert D. McBane, Director Vascular Medicine Division, Professor of Medicine, Mayo Clinic
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-009022
Record Dates: First submitted 2018-06-05; First posted 2018-07-18 (Actual); Results first posted 2020-03-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Deep Vein Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — apixaban

STUDY DESIGN:
Intervention Model Description: Multicenter, randomized, double blind, placebo-controlled, superiority clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind, placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Apixaban (Active Comparator): Apixaban 5mg (10 mg twice daily for 7 days followed by 5 mg twice daily for 3 months).
  Interventions: Drug: Apixaban
- Placebo (Placebo Comparator): Patients will receive matching placebo.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Apixaban — Active anticoagulation with apixaban 10 mg twice daily for 7 days followed by 5 mg twice daily to complete a total of 3 months treatment.
  Other Names: Eliquis
  Arms: Apixaban
Other: Placebo — apixaban matching placebo 2 tablets twice daily for 7 days followed by one tablet twice daily to complete a total of 3 months.
  Arms: Placebo

SUMMARY:
The primary objective is to evaluate whether apixaban is more effective in treating patients with isolated calf vein thrombosis (DVT) than serial imaging of the DVT for preventing thrombus spread, pulmonary embolism (PE) and/or recurring DVTs.

DETAILED DESCRIPTION:
This is a randomized double-blind placebo controlled superiority clinical trial. Patients will be identified at the time of the diagnosis of acute calf deep vein thrombosis and approached at that time. If they agree they would be randomly assigned to placebo or apixaban treatment for three months. Along with this they will also undergo repeat ultrasounds at 7, 14, and 90 days along with telephone follow-up at 30 and 60 days.

ELIGIBILITY:
Inclusion Criteria

1. Age range: ≥ 18 years.
2. Both males and females
3. Confirmed acute calf vein thrombosis confined to either the deep (posterior tibial, anterior tibial, or peroneal) or muscular (gastrocnemius or soleal) veins.
4. Negative serum or urine pregnancy test done (within 2 weeks) prior to randomization, for women of childbearing potential only. Note: A woman of childbearing potential (WOCBP) is defined as any female who has experienced menarche and who has not undergone surgical sterilization (hysterectomy or bilateral oophorectomy) and is not postmenopausal. Menopause is defined as 12 months of amenorrhea in a woman over age 45 years in the absence of other biological or physiological causes.
5. Ability to provide written informed consent.

Exclusion criteria

1. Any of the following because this study involves an investigational agent whose genotoxic, mutagenic and teratogenic effects on the developing fetus and newborn are unknown:

   * Pregnant women
   * Nursing women
   * Men or women of childbearing potential who are unwilling to employ adequate contraception Note: Women of child bearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 33 days after finishing the last dose.

   Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s) plus 93 days after finishing the last dose.

   Azoospermic males and WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements. However they must still undergo pregnancy testing as described in this section.

   Note: Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of an unexpected pregnancy Investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective methods of contraception. Highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly.

   At a minimum, subjects must agree to the use of one method of highly effective contraception as listed below:

   HIGHLY EFFECTIVE METHODS OF CONTRACEPTION
   * Male condoms with spermicide
   * Hormonal methods of contraception including combined oral contraceptive pills, vaginal ring, injectables, implants and intrauterine devices (IUDs) such as Mirena® by WOCBP subject or male subject's WOCBP partner.
   * Female partners of male subjects participating in the study may use hormone based contraceptives as one of the acceptable methods of contraception since they will not be receiving study drug,
   * IUDs such as ParaGard®,
   * Tubal ligation
   * Vasectomy.
   * Complete Abstinence* *Complete abstinence is defined as complete avoidance of heterosexual intercourse and is an acceptable form of contraception for all study drugs. Acceptable alternate methods of highly effective contraception must be discussed in the event that the subject chooses to forego complete abstinence
2. Acute co-existing proximal DVT (popliteal, femoral, iliac veins or IVC), pulmonary embolism, splanchnic vein thrombosis, cerebral venous sinus thrombosis within the past 3 months for whom anticoagulation therapy is indicated.
3. Age < 18 years.
4. Continuous treatment with therapeutic anticoagulant for more than 72 hours pre-randomization.
5. Contraindication to anticoagulant therapy
6. Significant kidney disease. Creatinine clearance < 25 ml/min using the Cockcroft-Gault equation: glomerular filtration rate (GFR) = (140-age) * (Wt in kg) * (0.85 if female) / (72 * Cr). (within last four weeks)
7. Significant liver disease (e.g. acute hepatitis, chronic active hepatitis, cirrhosis) or alanine transaminase (ALT) (or AST) > 3 x upper limit of normal (ULN). (within last four weeks)
8. Platelet count < 50 x109/L.(within last four weeks)
9. Life expectancy < 12 months.
10. Current active bleeding.
11. Concomitant use of strong CYP3A4 inhibitors (e.g., HIV protease inhibitors, systemic ketoconazole) or strong CYP3A4 inducers like rifampicin.
12. Active cancer defined as any evidence of cancer on cross-sectional imaging or cancer treatments within the past 6 months (chemotherapy, radiation therapy or cancer related surgery).
13. . Anticipated need for urgent/emergent surgery or major invasive procedure.
14. Dual antiplatelet therapy (thienopyridine plus aspirin) and/or aspirin greater than 165 mg while on study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2019-02-19 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D McBane, Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic, Eau Claire, Wisconsin
  - Mayo Clinic, La Crosse, Wisconsin

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Apixaban | Placebo
Started | 2 | 3
Completed | 2 | 2
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Apixaban | Placebo | Total
Number analyzed (Participants) | 2 | 3 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 77 (9.9) | 60 (17.69) | 67.3 (16.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 0 | 2 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 2 | 3 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Experience a Composite Venous Thromboembolism (VTE) Event Within 3 Months
Description: The composite VTE event will include thrombus propagation either within the calf veins or into proximal deep veins (popliteal, femoral or iliac veins), symptomatic or incidental VTE recurrence or all-cause mortality within 3 months of therapy initiation. All suspected VTE events will be evaluated by a central, blinded, independent adjudication committee.
Time Frame: Within 3 months of therapy initiation
Population: Study terminated due to lack of subject enrollment. Data was not analyzed.
Arm/Group | Apixaban | Placebo
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Number of Subjects Who Experience Either Major Bleeding or Clinically Relevant Non-major Bleeding Within 3 Months
Description: Major bleeding is defined as overt bleeding plus a hemoglobin decrease of ≥ 2 g/dL or transfusion of ≥ 2 units of packed red blood cells, or bleeding at a critical site: intracranial, intraspinal, intraocular, retroperitoneal, pericardial intra-articular, intramuscular with compartment syndrome, or fatal bleeding.
  Clinically relevant non-major bleeding is defined as any overt, actionable sign of hemorrhage meeting at least one of the following criteria: (i) requiring nonsurgical, medical intervention by a healthcare professional, (ii) leading to hospitalization or increased level of care, or (iii) prompting evaluation.
  All patients who received at least one dose of study medication will be included in the safety analysis. All suspected bleeding events will be evaluated by a central, blinded, independent adjudication committee.
Time Frame: Within 3 months of therapy initiation
Population: Study terminate to due lack of subject enrollment. Data was not analyzed.
Arm/Group | Apixaban | Placebo
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Mean Time of Thrombus Propagation
Description: The timing of thrombus propagation for those individuals who have suffered such an event. The date of thrombus propagation confirmation will be compared to the date of the original Deep Vein Thrombosis (DVT) diagnosis for this purpose.
Time Frame: Within 3 months of therapy initiation
Population: Study terminated due to lack of subject enrollment. Data was not analyzed.
Arm/Group | Apixaban | Placebo
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Net Clinical Benefit or Harm for the Two Strategies
Description: The outcome of net clinical benefit or harm will be assessed as the composite of the primary efficacy outcome or the principal safety outcome up to day 90. The difference in the incidences of the combined endpoint at 3 months between treatment arms will be estimated and tested using a normal approximation of the binomial distribution. All tests will be conducted at the two-sided 0.05 significance level.
Time Frame: Within 3 months of therapy initiation.
Population: Study terminated to due lack of subject enrollment. Data was not analyzed.
Arm/Group | Apixaban | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected for approximately 3 mos post enrollment for each subject
Arm/Group | Apixaban | Placebo
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 2/2 | 0/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Apixaban (N=2) | Placebo (N=3)
Nose Bleed (Vascular disorders) | 2 (2) | 0 (0)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Study was terminated due to lack of subjects enrollment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-05-10): https://cdn.clinicaltrials.gov/large-docs/43/NCT03590743/Prot_SAP_000.pdf